CLINICAL TRIAL: NCT06079515
Title: Comparison of the Treatment Efficacy of Suprascapular Nerve Block and Intraarticular Shoulder Injection Techniques in Patients Diagnosed With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000000000000
Record Dates: First submitted 2023-09-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Adhesive Capsulitis; Shoulder Pain
Keywords: adhesive capsulitis; suprascapular nerve blockade; intra-articular shoulder injection
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: A total of 60 patients who met the criteria and agreed to participate in the trial were included in the study. The patients were randomized into two groups suprascapular nerve block (SSNB) and intra-articular injection (IAI) using the closed envelope method.
Who Masked: Investigator
Masking Description: close envelope method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ali Akdağ (Active Comparator): All injections were performed by him under the guidance of a Clarius portable USG device (L7 HD Linear Ultrasound Scanner). A total of 10 ml of a mixture of 1 ml of 40 mg triamcinolone acetonide (Kenakort-A ampoule) and 9 ml of 0.5% bupivacaine hydrochloride (Marcaine) was used in each injection.
  Interventions: Procedure: Suprascapular Nerve Block; Procedure: Intraarticular Shoulder Injection
- Muhammet Hüseyin Sarı (Experimental): Blind observer to injections
  Interventions: Procedure: Suprascapular Nerve Block; Procedure: Intraarticular Shoulder Injection

INTERVENTIONS:
Procedure: Suprascapular Nerve Block — SSNB group: The patients were asked to sit comfortably in the chair, and the transducer was placed on the spine of the scapula in the coronal plane and moved laterally to observe the supraspinatus notch and the suprascapular nerve. The injection mixture was applied in-plane with a 22-gauge, 90-mm needle on the suprascapular nerve, under the fascia of the supraspinatus muscle.
Procedure: Intraarticular Shoulder Injection — IAI group: The patients were asked to sit on the chair with their hands facing the opposite shoulder, and the transducer was placed slightly below the spina scapula. The humeral head was observed by moving laterally. The injection mixture was applied in-plane with a 22-gauge, 90-mm needle entering the skin at a 45-degree angle and applied to the joint space

SUMMARY:
Objective: We aim to compare the efficiency of the ultrasonography-guided suprascapular nerve block (SSNB) and ultrasonography-guided intra-articular shoulder injection (IAI) techniques in terms of pain and functional status in the treatment of adhesive capsulitis.

Design: 60 patients with adhesive capsulitis were divided into two groups: SSNB and IAI. Both groups received an injection of 1 ml of 40 mg of triamcinolone acetonide and 9 ml of 0.5% bupivacaine hydrochloride. The patients' Shoulder Pain and Disability Index (SPADI) scores, shoulder active and passive range of motions (ROM), and visual analog scale (VAS) scores were evaluated before and after the injection in the 1st week, 4th week, and 12th week.

DETAILED DESCRIPTION:
Materials and Methods

Calculation of the Sample Size

The sample size of our study was calculated based on assuming the power of the study to be 80% and a type 1 (α) error of 0.05 using the G-Power 3.1.9.4 program. The sample size was calculated as 24 patients for each group. Considering the possibility of being excluded from the study, it was planned to recruit 30 patients for each group.

Patient Selection and Randomization

Our study was conducted at the Physical Therapy and Rehabilitation outpatient clinic of Antalya Education and Research Hospital between March and October 2022. A total of 84 patients aged between 18 and 75 who were found to be in the adhesive phase of AC after a detailed physical examination by the clinician were screened.

Patients with bilateral symptoms, radicular or inflammatory pain, uncontrolled DM, superficial infection at the injection site, bleeding disorder, stroke, history of drug allergy, shoulder trauma in the last month, any steroid injection in the last 3 months, pregnant or postpartum patients, and patients who had previously received shoulder physical therapy were excluded from the study.

As a result, a total of 60 patients who met the criteria and agreed to participate in the trial were included in the study. The patients were randomized into two groups suprascapular nerve block (SSNB) and intra-articular injection (IAI) using the closed envelope method.

Each patient was informed about the course of the disease, possible side effects of injections, and complications. Written informed consent was obtained from each patient. This study was approved by the Local Ethics Committee and was conducted by the principles of the Declaration of Helsinki.

Interventions

All injections were performed by a physiatrist with 15 years of experience under the guidance of a Clarius portable USG device (L7 HD Linear Ultrasound Scanner). A total of 10 ml of a mixture of 1 ml of 40 mg triamcinolone acetonide (Kenakort-A ampoule) and 9 ml of 0.5% bupivacaine hydrochloride (Marcaine) was used in each injection.

SSNB group: The patients were asked to sit comfortably in the chair, and the transducer was placed on the spine of the scapula in the coronal plane and moved laterally to observe the supraspinatus notch and the suprascapular nerve. The injection mixture was applied in-plane with a 22-gauge, 90-mm needle on the suprascapular nerve, under the fascia of the supraspinatus muscle.

IAI group: The patients were asked to sit on the chair with their hands facing the opposite shoulder, and the transducer was placed slightly below the spina scapula. The humeral head was observed by moving laterally. The injection mixture was applied in-plane with a 22-gauge, 90-mm needle entering the skin at a 45-degree angle and applied to the joint space.

In addition, both groups were given a home exercise program consisting of shoulder range of motion exercises in all directions, especially posterior capsule stretching, isometric strengthening exercises, and Codman exercises.

Clinical Evaluation

The primary outcome measure of the study was the Shoulder Pain and Disability Index (SPADI), and the secondary outcome measures were the Visual Analog Scale (VAS) and ROM measures. SPADI is a self-assessment scale with Turkish validity and reliability, consisting of two parts and a total of 13 questions; each question is given a score between 0 and 10. 21,22 Pain, disability, and total scores between 0 and 100 are obtained by calculating the percentage of the score indicated by the patients. SPADI variables were recorded as pain (SPADI-P), disability (SPADI-D), and total (SPADI-T) scores. VAS scores were marked between 0 and 100 mm by the patients. 23 ROM measurements, including active and passive shoulder flexion, abduction, extension, internal rotation, and external rotation, were measured with a goniometer.

All outcome measures were evaluated by an injection-blind clinician. Outcomes were evaluated four times: pre-injection, post-injection week 1, week 4, and week 12. Information such as age, gender, duration of symptoms, additional disease, affected side, and dominant extremity was recorded before the intervention.

Statistical Analysis

Descriptive statistics are presented with frequency, percentage, mean, standard deviation, median, minimum, and maximum values. In the analysis of categorical data, Fisher's Exact Test (Fisher's Exact Test) was used if the percentage of cells with the expected value less than 5 was greater than 20%, and the Pearson Chi-Square Test was used if it was small. The assumption of normality was checked with the Shapiro-Wilk Test. In the analysis of the difference between the numerical data of the two groups, the Independent Samples T-Test was used when the data conformed to the normal distribution, and the Mann-Whitney U-Test was used when they did not. Repeated measures ANOVA analysis was applied to compare the pre-injection, post-injection week 1, week 4, and week 12 measurements of the continuous numbers of variables according to the SSNB and IAI groups. Since the VAS score did not provide a normal distribution, the SSNB and IAI groups were evaluated within themselves with the Friedman test. Analyzes were made with the SPSS 23.0 program. A P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 to 75
* Adhesive phase

Exclusion Criteria:

* Patients with bilateral symptoms
* Radicular or inflammatory pain
* Uncontrolled DM
* Superficial infection at the injection site
* Bleeding disorder
* Stroke
* History of drug allergy
* Shoulder trauma in the last month
* Any steroid injection in the last 3 months
* Pregnant or postpartum patients
* Patients who had previously received shoulder physical therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | pre-injection, post-injection week 1, week 4, and week 12
  SPADI is a self-assessment scale with Turkish validity and reliability, consisting of two parts and a total of 13 questions; each question is scored between 0 and 10. Pain, disability, and total scores between 0 and 100 are obtained by calculating the percentage of the score indicated by the patients. SPADI variables were recorded as pain (SPADI-P), disability (SPADI-D), and total (SPADI-T) scores.
  Min score: 0 Max score: 100

SECONDARY OUTCOMES:
Visual Analog Scale | pre-injection, post-injection week 1, week 4, and week 12
  VAS scores were marked between 0 and 100 mm by the patients
  Min score: 0 Max score: 100
Shoulder Range of Motion | pre-injection, post-injection week 1, week 4, and week 12
  ROM measurements, including active and passive shoulder flexion, abduction, extension, internal rotation, and external rotation, were measured with a goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Education and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided